CLINICAL TRIAL: NCT02489279
Title: Training Attentional Awareness and Control in Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Training Attentional Awareness and Control in ADHD
Acronym: SAC-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Think Now Incorporated (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gregory Simpson, Ph.D., Founder and Chief Scientific Officer, Think Now Incorporated
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNI-SAC-I; R43MH101924 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention deficit hyperactivity disorder.; Attention training; Mobile devices; Brain training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — M Phase Cell Cycle Checkpoints; Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active - SAC (Experimental): Behavioral learning by using the Sustained Attention Control (SAC) Method's mobile software to increase sustained attention skills and self-awareness of attention control.
  Interventions: Behavioral: Sustained Attention Control (SAC) Method
- Control - Scrabble (Active Comparator): Behavioral learning using the mobile software game "Scrabble" to exercise word processing and executive control functions.
  Interventions: Behavioral: Scrabble

INTERVENTIONS:
Behavioral: Sustained Attention Control (SAC) Method — Participants use the software for 5 minutes, 3 times per day, 5 days per week, for 10 weeks.
  Arms: Active - SAC
Behavioral: Scrabble — Participants use the software for 5 minutes, 3 times per day, 5 days per week, for 10 weeks.
  Arms: Control - Scrabble

SUMMARY:
The purpose of this study is to evaluate the effects of different types of cognitive training on attention in adults with Attention Deficit Hyperactivity Disorder (ADHD) using mobile software on personal mobile devices.

DETAILED DESCRIPTION:
Different types of software-based cognitive training are thought to impact attention via different mechanisms. This study examines the nature of the effects on sustained attention of two different types of mobile software based training. Because the nature of the training method is behavioral, the investigators can not divulge the differences in the training methods and their hypothesized differences in their impact on attention.

ELIGIBILITY:
Inclusion Criteria:

1. Meet established Diagnostic and Statistical Manual-5 (DSM-5) criteria for ADHD predominately inattentive or combined subtype with clinically significant levels of impairment, diagnosed by structured clinical interview, the Mini International Neuropsychiatric Interview, and corroborating information
2. Clinical Global Impression-Severity (CGI-S) score ≥ 4 for ADHD
3. No lifetime history of DSM-5 bipolar disorder, psychotic disorder, pervasive developmental disorder, obsessive-compulsive disorder, substance abuse, or substance dependence (except nicotine) as assessed with the Mini-International Neuropsychiatric Interview (MINI)
4. Able in the opinion of the investigator to complete all required study procedures.

Exclusion Criteria:

1. History of diagnosis of childhood disorder other than ADHD (e.g. autism, dyslexia)
2. History of any general medical condition likely to require chronic use of medication with identified Central Nervous System (CNS) effects suspected to alter cognitive performance
3. History of seizure disorder, brain tumor, other major neurological disorder or head injury resulting in loss of consciousness
4. Serious oxygen deprivation
5. Current psychopathology requiring ongoing treatment with antipsychotic medications, mood stabilizers, benzodiazepines, or anticonvulsants
6. Current untreated psychopathology which is rated to be primary in terms of severity (greater than ADHD severity)
7. Current treatment with guanfacine.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Cohen, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from university clinics, local clinics, private practice clinicians and Attention-Deficit Hyperactivity Disorder (ADHD) groups.
Pre-assignment Details: 107 participants were screened and diagnosed and met eligibility criteria to be assigned to treatment. Of these, 22 declined to participate in the treatment stating that they changed their minds and that the treatment and follow-up testing would take too much time, leaving 85 randomized and assigned to treatment.
Groups:
- Active: Behavioral learning by using the Sustained Attention Control (SAC) Method's mobile software to increase sustained attention skills and self-awareness of attention control.
  Participants use the software for 5 minutes, 3 times per day, 5 days per week, for 10 weeks.
- Control: Behavioral learning using the mobile software game "Scrabble" to exercise word processing and executive control functions.
  Participants in both groups are told that the study is assessing the impact on cognitive tests from exercising with games that include cognitive processing. Scrabble serves as an active control with similar face value, equivalent usage and experimenter contact.
  Participants use the software for 5 minutes, 3 times per day, 5 days per week, for 10 weeks.
Period: Overall Study
Arm/Group | Active | Control
Started | 44 | 41
Completed | 32 | 31
Not Completed | 12 | 10
Not completed — Lost to Follow-up | 12 | 10

BASELINE CHARACTERISTICS:
Population: The demographics are based on the participants who completed all aspects of the study and for whom all outcome measurements were obtained.
Groups:
- Active: Behavioral training with the Attentional Intelligence Method mobile software to increase sustained attention skills and self-awareness of attention control.
  Attentional Intelligence Method: Participants use the mobile software, Attentional Intelligence Method, on their mobile device to develop sustained attention control and executive control skills that provides self-awareness of attention control. Participants use the software for 5 minutes, 3 times per day, 5 days per week, for 10 weeks.
- Control: Behavioral training with the mobile software game "Scrabble" to increase concentration.
  Scrabble: Participants play Scrabble on their mobile device to develop concentration and executive control skills. They use the software for 5 minutes, 3 times per day, 5 days per week, for 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.5 (5.44) | 27 (5.95) | 25.75 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 9 | 17 | 26
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63
Estimated Intelligence Quotient (IQ) [Mean (Standard Deviation); unit: IQ units (typical range 40-160).] — Estimate of IQ based on the composite score of the Wechsler Abbreviated Scale of Intelligence (WASI-II).
  IQ units (typical range 40-160). | 109.8 (10.7) | 107 (12.1) | 108.4 (11.4)
Years of education [Mean (Standard Deviation); unit: Years] | 15.1 (1.5) | 15.4 (1.7) | 15.25 (1.6)
ADHD Type [Number; unit: participants] — The ADHD Type (Inattentive or Combined) is based on the clinical diagnosis using the Adult ADHD Self Report Scale and structured interview. Population: Data were missing from 3 participants, leaving a total of 60. The determination of ADHD Type breaks the Overall participants into two groups.
  participants
    Inattentive Type: number analyzed (Participants) | 30 | 30 | 60
    Inattentive Type | 19 | 22 | 41
    Combined Type: number analyzed (Participants) | 30 | 30 | 60
    Combined Type | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Conners Continuous Performance Test (CPT) RT Variability Scaled Score
Description: Change was calculated as the score after 10 weeks of treatment minus the pre-treatment score at Baseline. This is a computerized continuous performance task yielding a measure of reaction time (RT) variability over the duration of the task as an assessment of sustained attention control. Less variability in RT is a sign of better sustained attention control. The scaled scores are T Scores and the range is 0-100. Smaller values represent better performance (i.e. lower variability). Consequently, a negative difference value (Post-Pre) indicates improvement. This measure directly addresses the training target, inconsistent control of sustained attention (the variability in RT over time), and is highly correlated with ADHD.
Time Frame: Baseline and 10 weeks
Population: Completer analysis of all subjects for whom Conners CPT RT Variability was measured at Baseline and after completing 10 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active - SAC | Control - Scrabble
Number analyzed (Participants) | 29 | 30
score on a scale | -6.65 (13.75) | 1.84 (14.80)
Statistical Analysis 1: Comparison: Active - SAC vs Control - Scrabble; We used a General Linear Model (GLM) with time (Baseline and 10 Weeks) as the within subjects factor, experimental group (Active and Control) as the between subjects factor, and a group by time interaction to test for differential treatment effects. We report the Group x Time interaction; Test type: Superiority; p = 0.026, GLM with repeated measures ANOVA
Statistical Analysis 2: Comparison: Active - SAC; We then examined the within-subjects factor of Time (Post-Treatment (10 week measure) - Baseline), for each Group, using a 1-tailed t test; Test type: Superiority; p = 0.0075, t-test, 1 sided
Statistical Analysis 3: Comparison: Control - Scrabble; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.25, t-test, 1 sided

2. Primary Outcome: Change From Baseline in Nelson-Denny Reading Test - Comprehension Score
Description: Change was calculated as the score after 10 weeks of treatment minus the pre-treatment score at Baseline. The Nelson Denny Reading Comprehension test is a time-limited (20-minute) measure of an important daily life activity that is impaired in ADHD, and impacted by poor sustained attention. The score range is from 0-76 with larger values representing better performance. A larger positive difference value (Post- Pre) indicates an improvement in reading comprehension.
Time Frame: Baseline and 10 weeks
Population: Completer analysis of all subjects for whom Nelson-Denny Reading Comprehension was measured at Baseline and after completing 10 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active - SAC | Control - Scrabble
Number analyzed (Participants) | 25 | 23
score on a scale | 7.36 (10.26) | 1.04 (6.09)
Statistical Analysis 1: Comparison: Active - SAC vs Control - Scrabble; We used a GLM with time (Baseline and 10 Weeks) as the within subjects factor, experimental group (Active and Control) as the between subjects factor, and a group by time interaction to test for differential treatment effects. We report the Group x Time interaction; Test type: Superiority; p = 0.014, GLM with repeated measures ANOVA
Statistical Analysis 2: Comparison: Active - SAC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0005, t-test, 1 sided
Statistical Analysis 3: Comparison: Control - Scrabble; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.21, t-test, 1 sided

3. Secondary Outcome: Change From Baseline in Adult Attention-Deficit Hyperactivity Disorder Self-Report Scale (ASRS) - Inattentive Subscale
Description: Change was calculated as the score after 10 weeks of treatment minus the pre-treatment score at Baseline. The ASRS is a scale to evaluate ADHD symptoms in adults. The Inattentive Symptoms Subscale range = 0-36. Higher values are worse. Consequently, a negative difference value indicates improvement.
Time Frame: Baseline and 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active - SAC | Control - Scrabble
Number analyzed (Participants) | 28 | 30
units on a scale | -3.29 (5.34) | -4.17 (4.67)
Statistical Analysis 1: Comparison: Active - SAC vs Control - Scrabble; We used a GLM with time (Baseline and 10 Weeks) as the within subjects factor, experimental group (Active and Control) as the between subjects factor, and a group by time interaction to test for differential treatment effects. We report only a main effect of Time; Test type: Superiority; p = 0.000001, GLM with repeated measures ANOVA

4. Secondary Outcome: Change From Baseline in Adult Attention-Deficit Hyperactivity Disorder Self-Report Scale (ASRS) - Hyperactive Subscale
Description: Change was calculated as the score after 10 weeks of treatment minus the pre-treatment score at Baseline. The ASRS is a scale to evaluate ADHD symptoms in adults. The Hyperactive Symptoms Subscale range = 0-36. Higher values are worse. Consequently, a negative difference value indicates improvement.
Time Frame: Baseline and 10 weeks
Population: Completer analysis of all subjects for whom ASRS was measured at Baseline and after completing 10 weeks of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active - SAC | Control - Scrabble
Number analyzed (Participants) | 28 | 30
units on a scale | -2.54 (5.34) | -3.13 (5.42)
Statistical Analysis 1: Comparison: Active - SAC vs Control - Scrabble; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.00018, GLM with repeated measures ANOVA

ADVERSE EVENTS:
Time Frame: 10 weeks from Baseline.
Description: The treatment and assessment methods have no known risks.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes